CLINICAL TRIAL: NCT07400848
Title: Clinical Laboratory Evaluation, Assessment of Symptoms and Recovery in Patients With Post-COVID-19-Vaccination Syndrome
Acronym: CLEAR
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: private practice Cell-Re-Active-Training in Bern (Unknown); Post-Vakzin-Syndrom Schweiz (Unknown); Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01382
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Post-Acute COVID-19 Vaccination Syndrome; Postviral Fatigue
Keywords: Vaccine-Related Adverse Event; Endothelial Dysfunction; Coagulation Abnormalities; Inflammation; Cytokines; Patient-Reported Outcomes; Symptom Burden; Disease Trajectory; Reactive Hyperemia Index
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-Acute COVID-19 Vaccination Syndrome Patients
  Interventions: Diagnostic Test: Blood sampling and analysis; Other: The continuous Reactive Hyperemia Index (InRHI) measured by EndoPAT
- Healthy controls: Matched (similar age (±10 years) and sex)
  Interventions: Diagnostic Test: Blood sampling and analysis; Other: The continuous Reactive Hyperemia Index (InRHI) measured by EndoPAT

INTERVENTIONS:
Diagnostic Test: Blood sampling and analysis — Blood sampling to analyze:
  1. Routine laboratory diagnostics including complete blood count, coagulation and inflammation markers (e.g., fibrinogen, von Willebrand Factor, D-dimer, Factor VIII, hsCRP, Troponin-T, NT-proBNP
  2. Platelet function analysis using the Multiplate Analyzer (ADPtest, ASPItest, TRAPtest)
  3. Blood morphology assessment using real-time confocal microscopy
  4. Endothelial activation (Syndecan-1, ICAM-1, PAI-1/tPA complex, Heparan sulfate)
  5. Complement activation (sC5b-9)
Other: The continuous Reactive Hyperemia Index (InRHI) measured by EndoPAT — To assess endothelial function, participants undergo a non-invasive measurement using the EndoPAT device. This system evaluates vascular reactivity by continuously recording the peripheral arterial tone (PAT) signal via pneumatic finger probes placed on both index fingers. The total duration of the measurement is approximately 17 minutes. During the first 6 minutes, the baseline vascular tone is recorded at rest. This is followed by a 5-minute arterial occlusion phase, during which a blood pressure cuff on one arm (typically the non-dominant arm) is inflated to suprasystolic pressure to temporarily interrupt arterial blood flow. After the cuff is released, the reactive hyperemia response is recorded for an additional 6 minutes to assess endothelial-dependent vasodilation. The procedure is painless and well-tolerated. Participants may experience a mild tingling sensation in the occluded arm during the occlusion phase. No adverse effects are expected.

SUMMARY:
Some people report persistent health problems after receiving the COVID-19 vaccine. These symptoms persist well beyond typical short-term vaccine side effects and are not attributable to any other known medical conditions. This condition is known as Post-Acute COVID-19 Vaccination Syndrome (PACVS). Symptoms can persist for months and affect several organ systems, causing issues such as fatigue, heart-related problems, neurological difficulties, and decreases in both physical ability and mental performance. PACVS shows similarities to Post-Acute COVID-19 syndrome (PACS) and myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS).

The biological processes that cause PACVS are still not fully understood. Recent research indicates that endothelial dysfunction, abnormalities in blood coagulation, and persistent inflammatory responses may contribute significantly to this process. However, it remains unclear how symptoms develop over time, which biological markers are associated with disease severity, and how these findings could support diagnosis and future treatment strategies.

The CLEAR study is an observational research project designed to address these knowledge gaps by systematically documenting symptoms over time and investigating potential biological correlates in individuals affected by PACVS. The study consists of three complementary subprojects.

The PROGRESS subproject aims to assess symptom burden, disease course, and patient-reported treatment experiences over an eight-month period using standardized questionnaires completed by participants.

The ENDOCLOT subproject investigates whether individuals with PACVS show objective signs of endothelial dysfunction, abnormalities in blood clotting, and markers of systemic inflammation. Endothelial function will be evaluated through non-invasive vascular reactivity tests (EndoPAT), microscopic examination of blood cells, standardized platelet function assessments, and standard laboratory diagnostics. It further explores the correlation between these biological parameters and clinical symptom trajectories identified in PROGRESS.

The REAL subproject examines the role of endothelial activation and the release of inflammatory signaling molecules (cytokines) in the development and persistence of PACVS.

The main hypothesis of the CLEAR study is that PACVS is associated with measurable endothelial dysfunction, inflammatory activation, and coagulation abnormalities, and that these biological changes are related to symptom severity and persistence over time. By combining longitudinal symptom assessment with biological measurements, this study aims to improve understanding of PACVS and support the development of better diagnostic and therapeutic approaches in the future.

ELIGIBILITY:
General Criteria (apply to all study parts: PROGRESS, ENDOCLOT, REAL, patients and matched healthy controls)

Inclusion Criteria

1. Age ≥ 18 years
2. Sufficient knowledge of German to complete study-related questionnaires and procedures

Exclusion Criteria

1. Severe cognitive, physical impairment or psychiatric conditions impeding participation
2. Active oncological disease or immunosuppressive
3. Known pregnancy at the time of enrolment

PROGRESS (patients only)

Inclusion Criteria

1. Coded participation with online consent confirmation
2. Self-reported onset of persistent symptoms temporally associated with a COVID-19 vaccination
3. Willingness and ability to participate in the 8-month follow-up period

Exclusion Criteria

1. No specific exclusion criteria for this part

ENDOCLOT and REAL (patients and matched healthy controls)

Inclusion Criteria

1. Signed informed consent form
2. For patients:

   1. Receipt of at least one COVID-19 vaccination
   2. Onset of new, otherwise unexplained symptoms within 0-14 days after vaccination
   3. Persistence of symptoms for at least 6 months following vaccination
   4. Selection is based on a diagnosis of ME/CFS according to the Canadian Consensus Criteria (CCC) and PEM.

2. For controls: History of COVID-19 vaccination without persistent adverse effects; age (+/- 10 years), and sex match to a corresponding case

Exclusion Criteria (patients and matched healthy controls)

1. Clinically suspected or laboratory confirmed SARS-CoV-2 infection after vaccination or temporally related to symptom onset.
2. Concurrent pre-existing Long COVID symptoms, obtained from the patient´s history
3. Any self-reported or uncertain history of an acute infectious event (including mild or subclinical infections) in temporal proximity to COVID-19 vaccination
4. Known pre-existing medical conditions or ongoing medications that could plausibly explain the reported symptoms (e.g., preexisting ME/CFS, POTS, fibromyalgia, small-fiberneuropathy, autoimmune disease with systemic involvement or other chronic multisystemic dysautonomia syndromes)
5. Use of long-term, high-dose anti-inflammatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Progress:The study aims to enrol approximately 150-200 adults (≥18 years) who report persistent and severe symptoms following COVID-19 vaccination.
  Endoclot/Real: The study includes 40 individuals with suspected PACVS who meet criteria for ME/CFS and PEM, as identified through the PROGRESS subproject. Each patient is matched with a healthy control of similar age (±10 years) and sex. Control participants must have received a COVID-19 vaccination but report no persistent adverse effects and no chronic illness.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Self-reported health status (EQ-VAS) | From enrollment to baseline assessment (T0)
  Self-reported overall health status measured using the EuroQoL Visual Analogue Scale (EQ-VAS), ranging from 0 to 100, with higher scores indicating better perceived health status.
Health-related quality of life (EQ-5D-5L index score) | From enrollment to baseline assessment T0
  Health-related quality of life assessed using the EuroQoL EQ-5D-5L index score, typically ranging from values below 0 (health states worse than death) to 1, with higher scores indicating better health-related quality of life.
Reactive Hyperemia Index (lnRHI) | From enrollment to the day of examination, estimated to occur within 14 days after enrollment.
  Continuous Reactive Hyperemia Index measured using EndoPAT; noting that values ≤0.51 indicating dysfunction

SECONDARY OUTCOMES:
Change in self-reported health status (EQ-VAS) | During follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks; T2) after enrollment.
  Self-reported health status measured using the EQ-VAS, ranging from 0 to 100, with higher scores indicating better perceived health status.
Change in health-related quality of life (EQ-5D-5L index score) | During follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Health-related quality of life measured using the EQ-5D-5L index score; higher scores indicate better quality of life.
Functional impairment (Bell Disability Scale) | From enrollment to baseline assessment (T0), and during follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Functional impairment assessed using the Bell Disability Scale, ranging from 0 to 100, with lower scores indicating greater disability.
ME/CFS symptom severity (Canadian Consensus Criteria) | From enrollment to baseline assessment (T0), and during follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Assessment of ME/CFS symptom severity, including fatigue, post-exertional malaise, unrefreshing sleep, pain, cognitive/neurological impairments, and autonomic, neuroendocrine, or immune manifestations. Symptoms are rated on a standardized scale, with higher scores indicating greater symptom severity and functional impairment.
Presence of post-exertional malaise (PEM) | From enrollment to baseline assessment (T0), and during follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Presence of post-exertional malaise assessed using a standardized PEM screening instrument (binary outcome: present/absent whereby at least one of the answer is indicated with a frequency and severity of ≥ 2. )
Functional capacity (FUNCAP55) | From enrollment to baseline assessment (T0), and during follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Functional capacity assessed using the FUNCAP55 screening instrument; higher scores indicate better functional capacity.
Reported treatments and medications | From enrollment to baseline assessment (T0), and during follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Self-reported past and current treatments and medications used by participants.
Self-reported treatment effects and side effects | From enrollment to baseline assessment (T0), and during follow-up at approximately 4 months (±2 weeks, T1) and 8 months (±2 weeks, T2) after enrollment.
  Participant-reported perceived treatment effects and adverse effects.
Platelet reactivity (ADPtest AUC) | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Platelet aggregation measured using Multiplate analyzer (ADPtest), reported as area under the curve (AUC); higher values indicate increased platelet reactivity.
Platelet reactivity (ASPItest AUC) | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Platelet aggregation measured using Multiplate analyzer (ASPItest), reported as area under the curve (AUC); higher values indicate increased platelet reactivity.
Platelet reactivity (TRAPtest AUC) | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Platelet aggregation measured using Multiplate analyzer (TRAPtest), reported as area under the curve (AUC); higher values indicate increased platelet reactivity.
High-sensitivity C-reactive protein (hs-CRP) level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Serum hs-CRP concentration; higher levels indicate increased systemic inflammation
Fibrinogen level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma fibrinogen concentration; higher levels indicate increased coagulation activity
D-dimer level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma D-dimer concentration; higher levels indicate increased fibrin turnover
von Willebrand factor level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma von Willebrand factor concentration; higher levels indicate endothelial activation.
Factor VIII activity | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma Factor VIII activity; higher activity indicates increased coagulation potential.
Troponin T (high sensitivity) | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  High-sensitivity cardiac troponin T concentration; higher levels indicate myocardial injury.
NT-proBNP level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma NT-proBNP concentration; higher levels indicate cardiac strain.
Blood cell morphology | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Microscopic assessment of leukocyte count and platelet and erythrocyte morphology.
Syndecan-1 level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma Syndecan-1 concentration; higher levels indicate increased endothelial activation.
ICAM-1 level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma ICAM-1 concentration; higher levels indicate endothelial activation.
PAI-1/tPA complex level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma PAI-1/tPA complex concentration; higher levels indicate impaired fibrinolysis.
Heparan sulfate level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma heparan sulfate concentration; higher levels indicate glycocalyx degradation.
Terminal complement complex (sC5b-9) level | From enrollment to the day of blood sampling, estimated to occur within 14 days after enrollment.
  Plasma sC5b-9 concentration; higher levels indicate complement activation.

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Schmidt, Prof. Dr., Principal Investigator — Institute of Sport Science, University of Bern, Switzerland; Dieter Thommen, Dr.med., Principal Investigator — Praxis für Cell-Re-Active-Training, Bern, Switzerland
Locations (1):
- Institute of Sport Science, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No